CLINICAL TRIAL: NCT04715607
Title: Comparison of Detection Rate of SARS-CoV-2 in Saliva, Oropharyngeal and Nasopharyngeal Specimens in a Public COVID-19 Test Setting
Brief Title: COVID-19: SARS-CoV-2 Detection in Saliva, Oropharyngeal and Nasopharyngeal Specimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Hvidovre University Hospital (Other); Region Hovedstadens Apotek (Other Government)
Responsible Party: Principal Investigator, Tobias Todsen, MD, PhD, Assistant professor Tobias Todsen, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2021-01
Record Dates: First submitted 2021-01-12; First posted 2021-01-20 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV Infection; Covid19; Coronavirus
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: All participants will have Saliva collected and recieve nasopharyngeal swabs and oropharyngeal swabs for SARS-COV2. To avoid systematic bias we plan to randomize the sequence of testing.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nasopharyngeal swab, oropharyngeal swab, and salvia collection (Active Comparator): The participants will first be tested with nasopharyngeal swabs followed by oropharyngeal swab and saliva collection.
  The collection material, virus transport medium and laboratory equipment for each method is the same in both arms
  Interventions: Diagnostic Test: Sequence of testing.
- Oropharyngeal swab, salvia collection, and nasopharyngeal swab (Active Comparator): The participants will first be tested with oropharyngeal swabs followed by saliva collection and nasopharyngeal swab.
  The collection material, virus transport medium and laboratory equipment for each method is the same in both arms
  Interventions: Diagnostic Test: Sequence of testing.
- Salvia collection, nasopharyngeal swab, and oropharyngeal swab (Active Comparator): The participants will first be tested with saliva collection followed by nasopharyngeal swab and oropharyngeal swabs.
  The collection material, virus transport medium and laboratory equipment for each method is the same in both arms
  Interventions: Diagnostic Test: Sequence of testing.

INTERVENTIONS:
Diagnostic Test: Sequence of testing. — The participants will be tested in the following sequences of sampling technique: (1) nasopharyngeal swab, oropharyngeal swab, and salvia collection OR (2) oropharyngeal swab, salvia collection, and nasopharyngeal swab OR (3) salvia collection, nasopharyngeal swab, and oropharyngeal swab. Only the sequence is different in the different arm, while the sampling technique for each method is the same in all arms.

SUMMARY:
The aim of this study is to compare the SARS-CoV-2 detection rate using either a Saliva, oropharyngeal swabs or nasopharyngeal swab method for specimen collection.

DETAILED DESCRIPTION:
The reference test to evaluate patients with suspected respiratory infection caused by virus is a real-time reverse transcription-polymerase chain reaction (RT-PCR) from a nasopharyngeal swab (NPS). However, other specimen collection methods like oropharyngeal swabs (OPS) and a saliva specimen collection have also been accepted by the Centers for Disease Control and Prevention for SARS-CoV-2 testing during the current coronavirus disease 19 (COVID-19) pandemic. It is unclear how much the SARS-CoV-2 detection rate differs when using different sampling methods and the aim of this study is to compare the expected COVID-19 detection rate using saliva, oropharyngeal swabs or nasopharyngeal swab in a public setting.

We, therefore, aim to investigate the detection rate of SARS-CoV-2 in Saliva, oropharyngeal swab, and nasopharyngeal swab specimen samples collected in symptomatic and non-symptomatic individuals tested for COVID-19 in a public test center during the COVID-19 pandemic.

Individuals referred for outpatient COVID-19 testing center will be invited to participate in a prospective clinical study. They will have saliva, OPS, and NPS specimen collection performed at the same time and analyzed separately for SARS-CoV-2. The rate for SARS-CoV-2 detection in saliva, OPS, and NPS will be compared using a logistic regression mixed-effect analysis. A Sample Size Calculation estimated that a sample of 18,000 participants would be needed for the trial with 80% power at a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* volunteers, who are attending the COVID-19 test facilities to obtain a RT-PCR test.
* oral and written informed consent to participate before entering the study.

Exclusion Criteria:

* Failure to understand and provide informed consent.
* Neck breathers (tracheostomy/laryngectomy patients) or other nasopharyngeal or oropharyngeal anomalies that do not allow for sampling using swabs.

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 27947 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 detection rates for oropharyngeal swabs (OPS) compared with nasopharyngeal swabs and saliva collection. | 48 hours after testing
  Due to the high specificity of RT-PCR, we will define a participant with an RT-PCR positive result from either Saliva, OPS or NPS as having a COVID-19 infection. The combined Saliva/OPS/NPS result will therefore be used as the diagnostic reference standard to calculate the sensitivity for the Saliva, OPS and NPS tests.

SECONDARY OUTCOMES:
SARS-CoV-2 RT-PCR cycle threshold (Ct) values | 48 hours after testing
  Ct values are compared between testing methods
OPS, NPS and saliva test discomfort and likelihood to get retested | immediately after testing (10 minutes)
  Discomfort scores (1-10) and likelihood to get retested are compared between testing methods
Ratio of mutations in SARS-CoV-2 | 48 hours after testing
  Detection rate of any mutations in SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Todsen, MD, PhD, Principal Investigator — Department of Otorhinolaryngology, Head and Neck Surgery and Audiology, Rigshospitalet; Nikolai Kirkby, MD, PhD, Study Director — Department of Clinical Microbiology, Rigshospitalet
Locations (1):
- Valby COVID-19 teststed, Copenhagen, Valby, Denmark

REFERENCES:
- [Derived] Todsen T, Tolsgaard MG, Benfield T, Folke F, Jakobsen KK, Gredal NT, Ersboll AK, von Buchwald C, Kirkby N. Higher SARS-CoV-2 detection of oropharyngeal compared with nasopharyngeal or saliva specimen for molecular testing: a multicentre randomised comparative accuracy study. Thorax. 2023 Oct;78(10):1028-1034. doi: 10.1136/thorax-2022-219599. Epub 2023 May 19. PMID 37208187
- [Derived] Todsen T, Tolsgaard M, Folke F, Jakobsen KK, Ersboll AK, Benfield T, von Buchwald C, Kirkby N. SARS-CoV-2 in saliva, oropharyngeal and nasopharyngeal specimens. Dan Med J. 2021 Apr 7;68(5):A01210087. PMID 33832565